CLINICAL TRIAL: NCT07387445
Title: Time Restricted Eating During Chemotherapy for Breast Cancer
Brief Title: A Multi-site Pilot Trial of Time Restircted Eating During Chemotheraply for Breast Cancer.
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Kelsey Nicole Dipman Gabel, Assistant Professor, University of Illinois at Chicago
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Study2021-0974
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer Early Stage Breast Cancer (Stage 1-3); Breast Neoplasm Female; Breast Cancer
Keywords: breast cancer; fasting; intermittent fasting; time restricted eating; chemotherapy initiation
MeSH Terms: conditions — Breast Neoplasms; Fasting; Intermittent Fasting

STUDY DESIGN:
Intervention Model Description: A 24-week open-label controlled trial will be conducted. Forty women with stage I-IV breast cancer initiating chemotherapy will be recruited. Women will be assigned to 8-h TRE (self-selected start at 10am, 11am, or 12pm) ad-libitum eating during a 24-week self-selected 8 hour eating window and fasting 16- hours daily, or standard care for 24 weeks.
Who Masked: Outcomes Assessor
Masking Description: data collectors and sample analysis will be blinded to arm allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care control (No Intervention): Participants assigned to standard care will follow the recommendations by American Association for Cancer Research and the American Cancer Society.
- 8-h TRE (Experimental): Participants assigned to this arm will follow the 8-h TRE protocol. Participants will consume food ad libitum (no calorie or food restrictions) during a self-selected 8-h eating window (beginning at 10:00 am, 11:00am, or 12:00 pm) and fasting for 16 hours daily. They will follow this same eating pattern for the length of the intervention. Calorie free drinks such as water, black coffee, and diet soda, are permitted during the fasting period. The eating window will allow for a typical breakfast/lunch/dinner eating pattern.
  Interventions: Behavioral: Time restricted eating

INTERVENTIONS:
Behavioral: Time restricted eating — Participants assigned to this arm will follow the 8-h TRE protocol. Participants will consume food ad libitum (no calorie or food restrictions) during a self-selected 8-h eating window (beginning at 10:00 am, 11:00am, or 12:00 pm) and fasting for 16 hours daily. They will follow this same eating pattern for the length of the intervention. Calorie free drinks such as water, black coffee, and diet soda, are permitted during the fasting period. The eating window will allow for a typical breakfast/lunch/dinner eating pattern.
  Other Names: TRE
  Arms: 8-h TRE

SUMMARY:
This study is being done to better understand how time restricted eating (eating all food in an 8 hour window) can help a person receiving chemotherapy treatment for breast cancer, stages I-IV. We want to find out if time restricted is feasible and acceptable to individuals starting chemotherapy for breast cancer. We will test 3 different eating window options compared to a control group for 24 weeks.

DETAILED DESCRIPTION:
We know very little about how nutrition therapy can affect breast cancer treatment outcomes. Current standard care suggests enough daily calories and protein to maintain body weight and avoid muscle loss. However, this approach may be antiquated given weight gain is common during treatment and emerging pre-clinical and clinical evidence suggest that fasting during chemotherapy may improve clinical and patient-reported outcomes. For example, preliminary human trials examining the fasting mimicking diet (very low-calorie, low-protein diet 1-week per month) or short-term fasting (48-120 hours (h)), known as periodic fasting, surrounding chemotherapy may increase effectiveness of treatment and decrease side effects related to chemotherapy. Yet these diets have low adherence, side effects of their own, and may increase patient burden and decrease quality of life. In contrast, time restricted eating (TRE) is a form of intermittent fasting with high adherence that may have similar positive effects on treatment outcomes without the untoward side-effects. Moreover, TRE may have beneficial effects on glucose regulation and body composition (i.e., decreased weight and body fat gain) suggesting the potential importance of this regimen to breast cancer recurrence. TRE is extremely accessible with no calorie counting or financial burden to the patient, individuals just shorten their eating window daily.

We aim to test the feasibility and acceptability of 24-weeks of 8-h TRE among female breast cancer patients initiating chemotherapy. Additionally we will examine the reliminary effect of 8-h TRE on treatment outcomes, treatment related side-effects, and patient reported quality of life and fatigue. Exploratory outcomes will include glucose regulation, body weight, body composition, IGF-1, IGFBP3, SHBG, estradiol (e2), TNF-alpha, and hsCRP

ELIGIBILITY:
Inclusion Criteria:

* Age 25-99 at time of consent
* English language or Spanish language (based on availability of lab interpreters)
* ECOG 0 or 1
* Breast cancer to meet histologically confirmed Stage I-III or Stage IV with Medical Oncology approval.
* Demonstrates adequate organ function (absolute neutrophil count ≥ 1,500/μL).
* All screening labs to be obtained within 30 days prior to registration.
* Able to provide written informed consent and HIPAA authorization for release of personal health information, via an approved UIC Institutional Review Board (IRB) informed consent form and HIPAA authorization.
* Women of childbearing potential must not be pregnant or breast-feeding. A negative serum or urine pregnancy test is required per institutional practice guidelines.
* As determined at the discretion of the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study.

Exclusion Criteria:

* Women with type 1 or insulin dependent type 2 diabetes
* Women with BMI > 45kg/m2 and < 18.5 kg/m2
* Women who are pregnant or nursing. A negative serum or urine pregnancy test is required per institutional practice guidelines.
* Shift workers
* Women with a history of eating disorders
* Enrolled participants with a significant weight loss or weight gain within 3 months of the study (weight gain or loss >4kg)
* Uncontrolled HIV/AIDS or active viral hepatitis
* Any prior malignancy <5 years, chemotherapy within the last year or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of this investigational regimen, as determined by the treating medical oncologist.
* Breast cancer recurrence classified by the treating medical oncologist
* Any mental or medical condition that prevents the patient from giving informed consent or participating in the trial.
* Other major comorbidity, as determined by study PI
* Illicit drug use within previous 3 months or excessive use of alcohol (i.e., > 2 drinks/day)
* Currently participating in Weight Watcher's or another weight loss program, including weight loss medication such as GLP-1 medications.
* Myocardial infarction
* Congestive heart failure
* Chronic hepatitis
* Cirrhosis
* Chronic pancreatitis
* History of solid organ transplantation

Ages: 25 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment feasibility | 24 weeks
  women eligible and referred by staff to the research team. We will also track the number of referred women approached (by phone & in person) by our research team for screening/enrollment and the number of women who decline and their reasons for non-enrollment
TRE Acceptibility | 24 weeks
  attendance at study visits, completeness of data, and overall and treatment specific loss to follow-up/withdrawal will be closely monitored
TRE adherence | 24 weeks
  Diet adherence will be monitored either by patient reported start and stop times of food intake and diet pattern scoring and will be assessed by the study coordinator with a total score of 7 days per week followed by a post intervention qualitative survey.

SECONDARY OUTCOMES:
Quality of Life | 24 weeks
  QLQ-C30
Fatigue | 24 weeks
  The Functional assessment of Cancer therapy - fatigue
Treatment related side effects | 24 weeks
  Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events, PRO-CTCAE
Safety | 24 weeks
  CBC
Change in Insulin | 24 weeks
Change in glucose | 24 weeks
Change in HbA1c | 24 weeks
Change in TNF-alpha | 24 weeks
Change in body weight | 24 weeks
Change in fat mass | 24 weeks
Change in lean mass | 24 weeks
Change in visceral adiposity | 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided